CLINICAL TRIAL: NCT04911426
Title: Telehealth-Clinical Advocacy Project
Acronym: (T-CAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R21DA048232-02 (NIH); 5R21DA048232-02 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-06-03 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Substance Use
Keywords: Opioids; Telehealth; Police diversion program
MeSH Terms: conditions — Substance-Related Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The two-arm randomization has been discontinued with new consented participants joining the study in 2023.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment plus telehealth (Experimental): Individuals will receive telehealth support services, including seven brief motivational interviewing sessions, delivered by a licensed substance use counselor via live interactive video calls during the 12-week intervention.
  Interventions: Behavioral: Telehealth

INTERVENTIONS:
Behavioral: Telehealth — The telehealth intervention is delivered with an app developed for this research. The intervention features live video calling, messaging, appointment reminders; clinical support is provided by licensed clinicians.

SUMMARY:
The purpose of this study is to develop a clinical telehealth intervention and test the feasibility of integrating telehealth within a police opioid county diversion program.

DETAILED DESCRIPTION:
Participants in a police opioid diversion program will receive information about the research opportunity; those interested will be administered informed consent and randomized to either the (1) diversion program treatment as usual condition or (2) the enhanced condition, receiving the telehealth video call intervention with motivational interviewing and substance use treatment appointment reminders during the 12-week intervention. The study design has been modified to provide the enhanced condition with coaching and the T-CAP app to all individuals consented to the study beginning January 1, 2023.

ELIGIBILITY:
Inclusion Criteria:

Individuals interested in joining the study will be

* Enrolled in the A Way Out Opioid Diversion Program (ODP),
* At least 18 years of age,
* Able to speak and understand English,
* Have a history of opioid, alcohol, or other substance use within last 12 months,
* Be willing to provide the research team with access to treatment records,
* Have access to a phone, tablet or computer for the informed consent activity, and
* Have a mailing address to receive a study phone issued to consented participants

Exclusion Criteria:

Individuals not eligible for the study are

* Not currently enrolled in the A Way Out Opioid Diversion Program on the day of consent,
* Under the age of 18 on the day of consent,
* Unable to speak and understand English,
* Have a history of past opioid, alcohol, or other substance use longer than 12 months ago with no use of opioids in the last 12 months,
* Unwilling to authorize the research team to access treatment records,
* Without access to a phone, tablet or computer to complete the informed consent activity,
* Without a mailing address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Pankow, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Lake County Public Health Department, Waukegan, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Plus Telehealth
Started | 8
Completed | 4
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Overall consented sample is N=8. Two individuals did not participate in the telehealth intervention and have been excluded in the analysis dataset (N=6).
Arm/Group | Treatment Plus Telehealth
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Number of Participants Completing the Texas Christian University Drug Screen 5 Data [Number; unit: participants] — The Texas Christian University Drug Screen 5 (TCUDS 5) is a 19-question survey that captures substance use during the past 12 months. The instrument includes subscale that gauges the severity of drug use corresponding with the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria based on a single disorder measured on the following continuum from mild to severe: mild disorder (presence of 2-3 symptoms); moderate disorder (presence of 4-5 symptoms); and severe disorder: (presence of 6 or more symptoms). The total score range is 0 to 11. Population: The sample size at baseline (N=8) in the analysis reflects that number of participants in the group who experienced the telehealth plus coaching intervention (n=6) and participants (n=2) who did not receive the intervention.
  participants | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Received One or More Referrals During the 12-week Intervention.
Description: The number of participants who received one or more referrals to services made by the intervention coach. This measure is collected as evidence supporting participant utilization of the app and the coaching support model.
Time Frame: 12-week intervention period
Population: Six of eight consented participants (i.e., the intent-to-treat participants) completed calls with a coach, resulting in four participants (n=66.67%) who received referrals and two participants (n=33.33%) who did not receive a referral. The remaining two participants were not in the intent-to-treat group after randomization was discontinued.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Plus Telehealth
Number analyzed (Participants) | 6
Participants | 4

2. Primary Outcome: Texas Christian University Drug Screen 5 Severity Score From Baseline to Post Intervention at Week 12
Description: The Texas Christian University Drug Screen 5 is a 19-question survey that captures substance use during the past 12 months. Interpretation of the TCU Drug Screen 5 score for drug use severity corresponds with the Diagnostic and Statistical Manual of Mental Disorders 5 criteria for reporting three possible severity levels (mild, moderate, severe). A single level score is based on participant responses to 11 items (total range: 0 to 11) as such: the presence of 2 to 3 endorsed symptoms is scored as a mild disorder; 4 to 5 endorsed symptoms is scored as moderate disorder; and a severe disorder is scored with the presence of 6 or more symptoms of the 11 items; thus, more endorsed items means a more serious drug use problem.
Time Frame: Texas Christian University Drug Screen 5 data are reported for baseline and end-of-intervention at 12 weeks after consent.
Population: Four participants completed the Texas Christian University Drug Screen 5 at baseline and at the end of the intervention (12 weeks after consenting to the study).
Measure: Mean (Full Range); unit: score on a scale
Groups:
- T-CAP Study Sample: Participants completed baseline assessment (Time 1) and also completed the assessment at the end of 12 weeks (Time 3).
Arm/Group | T-CAP Study Sample
Number analyzed (Participants) | 4
score on a scale
  TCU Drug Screen Baseline scores | 9.25 [0 to 11]
  Post intervention TCU Drug Screen Scores | 9.75 [0 to 11]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of 3 months.
Description: Definitions are consistent with Clinical Trials.
Arm/Group | Treatment Plus Telehealth
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Plus Telehealth (N=8)
Kidney stones (General disorders) | 1 (1) — Participant reporting medical care for kidney stones. Participant confirmed that there was no inpatient care for this illness and no surgery needed.
Medical procedure (General disorders) | 1 (1) — Undetermined health issue reported by the participant that did not include an overnight hospital stay.

LIMITATIONS AND CAVEATS:
The T-CAP project explored the feasibility of implementing a telehealth model in a police diversion program that supports adults in recovery from opioid use disorder with treatment as an alternative to arrest. Inadequate data collection due to enrollment well below the target during the 2019 pandemic limits the ability to draw meaningful conclusions about the impact of the intervention to support people in recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT04911426/Prot_SAP_000.pdf